CLINICAL TRIAL: NCT06160596
Title: Analyzing and Solving Exceptional Long-term Survivors in Solid Tumors With Poor Prognosis: A 3 Cohorts Case Control Matched Study
Brief Title: Analyzing and Solving Exceptional Long-term Survivors in Solid Tumors With Poor Prognosis
Acronym: ROSALIND
Status: Recruiting | Type: Observational
Sponsor: Cure 51 (Other)
Collaborators: Gustave Roussy, Cancer Campus, Grand Paris (Other); Centre Leon Berard (Other); Vall d'Hebron Institute of Oncology (Other); Istituto Europeo di Oncologia (Other); Charite University, Berlin, Germany (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-A02541-42
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Pancreas Adenocarcinoma; Small-cell Lung Cancer; Glioblastoma, IDH-wildtype
MeSH Terms: conditions — Small Cell Lung Carcinoma; Glioblastoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Biopsies, surgical pieces, frozen plasma, blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- PDAC STAGE IV SURVIVORS & CONTROLS: Metastatic pancreatic ductal adenocarcinoma (PDAC) (Other histologies such as adenosquamous carcinoma, hepatoid carcinoma, anaplastic undifferentiated carcinoma and medullary carcinoma, acinar cell carcinoma, neuroendocrine tumors, Solid pseudopapillary neoplasm, Pancreatoblastoma, Serous cystadenocarcinoma are excluded)
  Interventions: Genetic: Long term survival multimodal analysis
- SMALL CELL LUNG CANCER EXTENSIVE STAGE SURVIVORS & CONTROLS: Extensive small cell lung cancer (SCLC) (Other histologies excluded: combined SCLC with some areas of non-small cell lung cancer (NSCLC), carcinoid tumors, typical and atypical, large cell neuroendocrine carcinoma of the lung).
  Interventions: Genetic: Long term survival multimodal analysis
- GLIOBLASTOMA SURVIVORS & CONTROLS: Glioblastoma (GBM) (IDH mutated excluded)
  Interventions: Genetic: Long term survival multimodal analysis

INTERVENTIONS:
Genetic: Long term survival multimodal analysis — * To describe global signatures (Digital histology, Radiomic, Genomic, Transcriptomic, Proteomic, (Epigenomic) and clinical signature) that are associated with a patient's unexpected survival compared to standard patients across three cohorts of solid tumors with unmet medical needs.
  * To describe global signatures in the overall population (pan-cohort).
  * To describe clinical, digital pathology, radiomic, genomic, transcriptomic, proteomic and epigenomic signatures associated with patients' unexpected survival compared to standard patients for each cohort and in all cohorts (pan-cohort)

SUMMARY:
This is a retrospective, exploratory, multi-center, translational, 3 cohorts case control matched study conducted in patients harboring a solid tumor with poor prognosis who presented a long-term (case) and standard (standard) survival.

Patients with:

* Cohort A: metastatic pancreatic ductal adenocarcinoma
* Cohort B: glioblastoma IDHwt
* Cohort C: extensive small cell lung cancer

This research aims to integrate data generated from clinical records, imaging, multi-omics and bioinformatics approaches to discriminate case and control and then to identify new therapeutic targets. Analyses will be performed depending on the tumor samples available with at least 3 omics levels and according to scientific advances; genomic, epigenomic, proteomics, metabolomics, transcriptomic, microbiomic.

DETAILED DESCRIPTION:
We propose for the first time to build a large collection of samples from unexpected survivors and controls with standard survival to identify biomarkers of resistance and/or survival which would help developing new cancer therapeutics. Biological samples and clinical records will be collected and then centralised to extract the data of any patients who have survived more than 5 years for the cohorts of PDAC and SCLC and more than 3 years for the cohort of GMB-IDHwt from the day of diagnosis. In addition to the clinical record of the patient describing his/her history (including multiscale imaging, pathology, biological sample analysis), we will collect every point of data possible with current technologies, such as multi-omics including genome, proteome, transcriptome, epigenomic, metabolome and microbiome. The data set of these multi-omic groups are combined and are complementary to identify a certain biological function and its cellular source. Such complementary effects and synergistic interactions between omic layers in the life course can only be captured by integrative study of multiple molecular layers. Artificial intelligence (AI), specifically machine learning algorithms, will also help to understand these multi-omics data. AI can also bring a new layer of biomarker discovery enabling the analysis of whole slide images of biopsies with computer vision and linking those biomarkers to the multi omics genomic features. After interpreting the comprehensive data with our set-up bioinformatics team in coordination with the various centres, we expect to find molecular signatures and consequently therapeutic approaches to address patients and physicians unmet needs.

ELIGIBILITY:
Inclusion Criteria:

FOR SURVIVORS

* To be eligible the exceptional survivor patients must fulfill the following inclusion criteria:

  1. Adult patient (≥18 years old at diagnosis).
  2. Three distinct cohorts, one of patients harbouring metastatic pancreatic ductal adenocarcinoma, glioblastoma IDHwt, extensive small cell lung cancer.
  3. Long-term survival is defined as an exceptionally long survival ≥ 5 years from stage IV diagnosis for PDAC, extensive SCLC, and ≥ 3 years for GBM-IDHwt.
  4. Availability of at least one block sample and associated clinical annotations with following characteristics:

     * One block sample must be of sufficient quality and in sufficient quantity to perform multi-omic analyses, according to requirements specified in Lab manual
     * Any treatment prior to sample acquisition must be reported - all treatments accepted (standard / targeted);
     * Samples should be at least 5 years old for PDAC and SCLC and 3 years old for GBM

For CONTROL GROUPS :

* To be eligible the control patients must fulfill the following inclusion criteria:

  1. ≥18 years old at diagnosis.
  2. Three distinct cohorts, one of patients suffering from metastatic pancreatic ductal adenocarcinoma, one for glioblastoma, one for extensive small cell lung cancer.
  3. Paired to long-term survivors as mentioned in the methodology section
  4. Death or median overall survival with a variation of 10% before of beyond as reported in pivotal clinical trials in the specific type disease
  5. Availability of at least one tumor sample and associated clinical annotations with following characteristics:

     * Sample must be of sufficient quality and in sufficient quantity to perform multi-omic analyses
     * Any treatment prior to sample acquisition must be reported (treatment-naive samples should be preferred) - all treatments accepted (standard / targeted).

     Exclusion Criteria for both groups :
* Patient must not be enrolled if he/she fulfils one of the following non-inclusion criteria:

  1. <18 years old at diagnosis.
  2. Hematological malignancy or solid tumors, which are not in the scope of tumor types, described in the inclusion criteria.
  3. Tumor sample not available or not reaching the required quality for multi-omic analyses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary and secondary care clinic, oncology centers
Sampling Method: Non-Probability Sample
Enrollment: 1020 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
EXCEPTIONAL SURVIVAL | 54 months
  In this study, the primary endpoint is the long survivorship status (Y/N). Prior to locking the database, a data review meeting will be planned to review individual data and validate the Statistical Analysis Plan (SAP).
  All the deviations from protocol definitions (if any) will be listed and defined as major or minor deviations in the SAP.

CONTACTS AND LOCATIONS:
Overall Officials: Julieta Rodriguez, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Gustave Roussy Cancer Campus, Grand Paris, Villejuif, France

IPD SHARING:
Plan to Share IPD: No
To be discussed internally and with the scientific advisory board later. All institutions providing patient data will have full access to multiomics sequencing raw data of their own patients for academic use.

REFERENCES:
- See also: corporate website of sponsor — http://www.cure51.com